CLINICAL TRIAL: NCT02520817
Title: Professor of Tropical Medicine
Brief Title: Antioxidants and Zinc Improving Minimal Hepatic Encephalopathy In Truck Drivers; a Pilot Study
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nasser Mousa, Professor of Tropical Medicine, Mansoura University
Other Study IDs: Nasser hamed ahmed Mousa
Record Dates: First submitted 2015-07-23; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: Antioxidants; Zinc; Truck drivers
MeSH Terms: interventions — gluconic acid; Vitamin A; Ascorbic Acid; Lactulose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Antioxidant supplementation and zinc plus Lactulose(Group A): Patients With MHE were assigned to receive zinc and antioxidant plus lactulose (group A)
  Interventions: Dietary Supplement: 175 mg zinc gluconate, 50000 IU vitamin A, 500 mg vitamin C and 100 mg vitamin E once daily plus lactulose; dose 30-60 ml/day for 3 months
- Lactulose only (Group B): Patients with MHE were assigned to receive lactulose oly (group B)
  Interventions: Dietary Supplement: Lactulose

INTERVENTIONS:
Dietary Supplement: 175 mg zinc gluconate, 50000 IU vitamin A, 500 mg vitamin C and 100 mg vitamin E once daily plus lactulose; dose 30-60 ml/day for 3 months
  Groups: Antioxidant supplementation and zinc plus Lactulose(Group A)
Dietary Supplement: Lactulose
  Groups: Lactulose only (Group B)

SUMMARY:
Minimal hepatic encephalopathy (MHE) can have a far-reaching impact on quality and ability to function in daily life and may progress to overt Hepatic Encephalopathy. Patients with MHE were missed in clinical follow up and are more exposure to work accident. The aim of the present study was to assess the effects of oral supplementation of antioxidant and zinc gluconate Versus Lactulose inTruck driver cirrhotic patients with MHE.

DETAILED DESCRIPTION:
The aim of the present study was to assess the effects of oral supplementation of antioxidant and zinc gluconate in patients with MHE. Zinc, may be considered as a cofactor of urea cycle enzymes, that deficient in cirrhotic patients; especially if associated, with malnutrition or encephalopathy . Zinc is essential for the synthesis of coenzymes that mediate biogenic amine synthesis and metabolism. Data from studies sustain that, there is a synergistic combined effect between systemic oxidative stress, and ammonia that is implicated in the pathogenesis of hepatic encephalopathy, so that the present study was designed to assess the effects of oral supplementation of antioxidant and zinc gluconate in cirrhotic Truck drivers patients with MHE.

A prospective randomized controlled study comparing the effect of zinc and antioxidant supplementation plus lactulose on MHE versus lactulose alone. Patients who were diagnosed as having MHE were randomly assigned either to receive zinc and antioxidant plus lactulose (group A) or lactulose alone (group B, the control). Patients in group A received 175 mg zinc gluconate, 50000 iu vitamin A, 500 mg vitamin C and 100 mg vitamin E once daily plus lactulose (30-60 ml in 2 or 3 divided doses), while patients in group B received 30-60 ml lactulose in 2 or 3 divided doses so that the patient passed 2-3 semi soft stools per day. The therapy was taken daily for 3 months or until the patients discontinued the study drugs for any reason (e.g. non compliance). All patients were followed up every month for treatment compliance and for development of any complications. The compliance with the therapy was assured primarily by ensuring increased stool frequency and a change to a softer consistency and by counting the number of bottles of lactulose consumed. None of the study, patients were specifically treated by other therapy for MHE within the study period (e.g. rifaximin).

ELIGIBILITY:
Inclusion Criteria:

* Truck drivers with liver cirrhosis and minimal hepatic encephalopathy.

Exclusion criteria:

* Overt hepatic encephalopathy.
* Sensory or motor deficits; neurological causes of impaired cognition
* Electrolyte imbalances (serum sodium level <125 mmol/L; serum calcium level >10 mg per /DL and potassium level <2.5 mmol/L)
* Ongoing systemic illnesses, intercurrent infection or active spontaneous bacterial peritonitis.
* Recent history (< 6 weeks) of alcohol intake.
* Patients on drugs affecting psychometric performances.
* Recent (<6 weeks) intake of antibiotics for gastrointestinal bleeding, history of shunt operation or trans jugular intrahepatic portosystemic shunt for portal hypertension.
* Chronic renal impairment (creatinine level >2.0 mg per/ DL.
* Patients with color blindness, mature cataract and diabetic retinopathy,
* Hepatocellular carcinoma, or other comorbidities such as congestive heart failure and pulmonary disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutive patients (truck drivers) with liver cirrhosis were screened for MHE. The patients attended the Tropical and Neurology Outpatient clinics in Mansoura university Hospital, Mansoura
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Neuropsychometric tests including number connection test-part A, digit symbol test and block-design test. | 3 months
Serum ammonia levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tropical Medicine Tropical Medicine, Principal Investigator — Tropical Medicine
Locations (1):
- Nasser H Mousa,MD,mousa_medic@yahoo.com. +201227029213, Al Mansurah, Egypt